CLINICAL TRIAL: NCT04343469
Title: Effects of Morbid Obesity and Bariatric Surgery on Brain Inflammation, Insulin Resistance and Activation of Central Reward System Studied Using PET- and MRI-imaging
Brief Title: Effects of Morbid Obesity and Bariatric Surgery on Brain Inflammation, and Activation of Central Reward System
Acronym: BARIBRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, Professor, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: T26/2019
Record Dates: First submitted 2019-10-07; First posted 2020-04-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Morbid Obesity
Keywords: positron emission tomography; magnetic resonance imaging; euglycaemic hyperinsulinemic clamp; astrogliosis; central inflammation; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Gliosis | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Obese and healthy ones are compared at baseline and obese are compered to healthy ones 6 months after bariatric surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric surgery (Active Comparator): The effect of bariatric surgery (RYGB or LSG) on central inflammation
  Interventions: Procedure: Bariatric Surgery (RYGB or LSG)
- No intervention (No Intervention): Healthy lean volunteers

INTERVENTIONS:
Procedure: Bariatric Surgery (RYGB or LSG) — Morbidly obese subjects will receive either RYGB or LSG, and the effect of bariatric surgery-induced weight loss on brain inflammation will be assessed
  Arms: Bariatric surgery

SUMMARY:
Background: The investigators have found that obesity and insulin resistance result in significantly increased brain insulin-stimulated glucose uptake, whereas in every other tissue glucose uptake is lower in the obese compared to lean individuals. One possible explanation to this could be central inflammation and activation of brain glial cells, which has been shown to occur in animal models of obesity.

Aims: The objective of this study is to investigate whether there is brain inflammation in human obesity, and whether weight loss following bariatric surgery decreases brain inflammation.

Methods: A total of 60 morbidly obese subjects, assigned for Roux-en-Y gastric bypass or for sleeve gastrectomy according to routine treatment protocols will be recruited for this study. A control group of 30 healthy subjects will also be recruited. The following studies will be performed to patients and healthy subjects: 1) structural MRI and MRS, 2) functional MRI, 3) PET imaging of cerebral inflammation and astrocyte activation using [11C]-PK11195, 4) measurement of whole-body and tissue insulin sensitivity by combining hyperinsulinemic, euglycemic clamp with [18F]-FDG-PET, 5) neuropsychological testing. The study procedures will be repeated for the morbidly obese 6 months postoperatively.

DETAILED DESCRIPTION:
This is a prospective study, where subjects for the morbidly obese group (N=60) will be recruited from the patients undergoing bariatric surgery according to normal treatment protocol and the bariatric procedure is decided on clinical data together with the bariatric surgeon and the patient. The morbidly obese patients are studied before and 6 months after bariatric surgery.

Results of obese are compared to results of healthy subjects (N=30), who are studied once.

MRI studies: Brain structural MRI and MRS Structural brain MRI will be performed to obtain anatomical reference. The MR part of a 3T PET-MR system will be used for the study . MR spectroscopy (MRS) will be used to determine levels of different metabolites.Brain activation studies (functional MRI) The aim of the fMRI is to assess how morbid obesity and weight loss influence the brain reward system in response to visual cues (not food related); resting state fMRI will also be performed.

Brain inflammation: [¹¹C]-PK11195 tracer with PET/CT is used to determine activation of glial cells, or inflammation, in the brain. After intravenous injection of 500 MBq [¹¹C]-PK11195, a 60-minute dynamic scan on the brain using the same PET/CT cameras will be performed. Both ROI- and SPM based statistics will be used in the statistical analyses.

Whole-body scan with [18F]-FDG and PET/CT during euglycemic hyperinsulinemia used to promote tissue glucose uptake and measure insulin sensitivity. After 60 minutes from the start of clamp, the subjects will be injected intravenously with 150 MBq of [18F]-fluorodeoxyglucose ([18F]-FDG) Thereafter [18F]-fluorodeoxyglucose uptake in the brain, abdomen, femoral region will be measured.

ELIGIBILITY:
For the morbidly obese subjects:

1. BMI 35.0-45.0 kg/m2, or BMI 32.0-45.0 kg/m2 and diagnosed diabetes
2. Eligible to bariatric surgery evaluated according to normal treatment paradigm

Exclusion Criteria:

1. Metal objects in the body (including pacemakers, metallic artificial valve prostheses, inner ear implants, surgical clips, braces, foreign fragments)
2. Previous participation in PET studies
3. Pregnancy
4. Poor compliance, alcohol or drug abuse
5. Weight over 150 kg or waist circumference over 150 cm
6. Diabetes with fasting glucose levels ≥7.0 mmol/L, or treatment with insulin
7. Any chronic disease, medication or condition that could create a hazard to subject safety, endanger study procedures or interfere with the interpretation of results.

For the lean control subjects:

Inclusion Criteria:

1. BMI 18-27 kg/m2
2. Fasting plasma glucose ≤6.1 mmol/L
3. Normal values in 2-hour oral glucose tolerance test

Exclusion Criteria:

1. Metal objects in the body (including pacemakers, metallic artificial valve prostheses, inner ear implants, surgical clips, braces, foreign fragments)
2. Previous participation in PET studies
3. Pregnancy
4. Poor compliance, alcohol or drug abuse
5. Smoking
6. History of eating disorders, drastic weight-gain or weight-loss
7. History of psychiatric disorders
8. Any chronic disease, medication or condition that could create a hazard to subject safety, endanger study procedures or interfere with the interpretation of results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Obese have brain inflammation compared to healthy ones | Both groups at baseline
  Brain PET-[11C]-PK11195 imaging study of obese and healthy lean ones
Bariatric surgery decreases brain inflammation in obesity | Baseline and 6 months after operation (obese group only)
  PK11195 imaging results are compared before and 6 months after bariatric surgery in obese group studied before and after bariatric surgery

SECONDARY OUTCOMES:
Tissue-specific and whole-body insulin sensitivity are decreased in obese | Baseline obese and leans
  Glucose uptakes are measured using PET imaging in obese and leans
Tissue-specific and whole-body glucose improves after bariatric surgery | PET imaging studies at baseline and 6 months after operation
  Comparison before and 6 months after surgery (obese group)
Brain neural activity decreased in obesity | Baseline obese and leans
  Comparison between obese and lean ones using fMRI
Brain neural activity improves after bariatric surgery | Baseline and 6 months after operation (obese group)
  Comparison between obese baseline and 6 months after operation
Brain metabolite concentrations are different in obese | Baseline obese and leans
  MRS studies for obese and lean ones at baseline are compared
Brain metabolite concentrations normalize after bariatric surgery | Baseline and 6 months postop (obese group)
  MRS studies for obese before and 6 months postop compared

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD, PhD, Principal Investigator — Turku UH
Locations (2):
- Finland (2):
  - Turku PET Centre, Turku
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No